CLINICAL TRIAL: NCT03414580
Title: Analysis of Volatile Organic Compounds in Exhaled Air in Patients With Inflammatory Bowel Disease Patients and Healthy Control
Brief Title: Analysis of Volatile Organic Compounds in the Exhaled Air in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, YooJin Lee, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2017-08-003
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Volatile Organic Compounds; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Volatile Organic Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ulcerative colitis: Patients with ulcerative colitis whose diagnosis had established on clinical, endoscopic, histologic, and/or radiological criteria. Breath sampling for volatile organic compounds will be analysed by gas chromatography-mass spectrometry.
  Interventions: Procedure: Breath sampling for volatile organic compounds
- Crohn's disease: Patients with crohn's disease whose diagnosis had established on clinical, endoscopic, histologic, and/or radiological criteria. Breath sampling for volatile organic compounds will be analysed by gas chromatography-mass spectrometry.
  Interventions: Procedure: Breath sampling for volatile organic compounds
- Healthy control: Subject with no intestinal symptoms or no known gastrointestinal disorders. Breath sampling for volatile organic compounds will be analysed by gas chromatography-mass spectrometry.
  Interventions: Procedure: Breath sampling for volatile organic compounds

INTERVENTIONS:
Procedure: Breath sampling for volatile organic compounds — Acquisition of exhaled breath sample in exhaled air to be analysed by gas chromatography-mass spectrometry

SUMMARY:
The availability of noninvasive biomarkers for diagnosis and stratification of inflammatory bowel disease (IBD) courses is lacking. Thus, the aim of this study is to evaluated the accuracy of exhaled breath volatile metabolite analysis on diagnosis and stratification of patients with inflammatory bowel disease.

DETAILED DESCRIPTION:
Background: The diagnosis and differentiation of inflammatory bowel diseases (IBD) is challenging due to the absence of a gold standard diagnostic modality for confirmation. Exhaled breath volatile metabolite analysis focusing on diagnosis and differentiation of IBD is a promising approach. Thus, the aim of this study is to evaluated the accuracy of exhaled breath volatile metabolite analysis for patients with inflammatory bowel disease.

Method: A single center, prospective study of diagnostic testing will be conducted, recruiting crohn's disease (CD), ulcerative colitis (UC), and healthy controls (HC). The exhaled breath volatile metabolite will be analyzed using gas chromatography/mass spectrometry (GC-MS). The informations of patient's disease location, disease activity, laboratory parameters and current medications will be collected to determine the feasibility of exhaled breath volatile metabolite analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Healthy controls who do not have any gastrointestinal disease or symptom

Exclusion Criteria:

* Pregnant or lactating woman
* Subjects who diagnosed liver cirrhosis, severe congestive heart failure, severe renal insufficiency, uncontrolled hypertension, endocrine disorder, metabolic disorder, prior malignancy, immune deficiency
* Subjects with mental retardation and cognitive impairment

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease visiting the Keimyung University Dong San Medical center will be eligible.
  Subject without any gastrointestinal disease or symptom will be eligible as healthy control group.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Volatile organic compounds differentiating the study groups | At the time of breath sampling
  Volatile organic compounds analysed by GC-MS between the study groups

SECONDARY OUTCOMES:
Volatile organic compounds differentiating the disease activity | At the time of breath sampling
  Volatile organic compounds analysed by GC-MS between the study groups

CONTACTS AND LOCATIONS:
Overall Officials: Yoo Jin Lee, Professor, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- KeimyungUniversity, Daegu, Jung-gu, South Korea